CLINICAL TRIAL: NCT00262483
Title: A Phase 2 Study of VX-950 in Combination With Peginterferon Alfa-2a (Pegasys®) and Ribavirin (Copegus®) in Subjects With Hepatitis C
Brief Title: Phase 2 Study of VX-950, Pegasys and Copegus in Hepatitis C
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Robert Kauffman M.D., Ph.D., Vertex Pharmaceuticals Incorporated
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: VX05-950-102
Record Dates: First submitted 2005-12-02; First posted 2005-12-06 (Estimated); Last update posted 2007-12-21 (Estimated); Status verified 2007-12

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — telaprevir; Ribavirin; peginterferon alfa-2a

INTERVENTIONS:
Drug: VX-950
Drug: ribavirin
Drug: peginterferon alfa-2a

SUMMARY:
To assess the safety of the combination of VX-950, Pegasys and Copegus in subjects with hepatitis C.

ELIGIBILITY:
Inclusion Criteria:

* Infected with hepatitis C virus

Exclusion Criteria:

* Contraindications to peginterferon or ribavirin therapy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12
Dates: Start 2005-12; Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Safety of triple combination therapy. | retrospective and prospective

SECONDARY OUTCOMES:
Pharmacokinetics of VX-950, peginterferon alfa-2a and ribavirin. | retrospective and prospective
Plasma HCV RNA levels | retrospective and prospective

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Vertex Pharmaceuticals Incorporated
Locations (2):
- Call for information, San Antonio, Texas, United States
- Call for information, Santurce, Puerto Rico